CLINICAL TRIAL: NCT06827184
Title: By Assessing the Continuous Respiratory Physiological Changes Through Prone Position, Determine the Optimal Duration for Prone Position
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 202310137DIND
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Distress Syndrome; Prone Position; Electrical Impedance Tomography
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Electrical Impedance Tomography — It utilizes electrical impedance tomography to analyze a series of physiological changes in the lungs following treatment

SUMMARY:
The prone position leads to a more homogeneous distribution of ventilation by inflation of collapsed alveoli and reduction in alveolar hyperinflation. By employing EIT, the study can obtain a thorough comprehension of the ongoing alterations in regional ventilation before and after adopting the prone position. It is also anticipated that there is an impact on inflammation biomarkers before and after the prone position. This assessment aids in determining the ideal duration for prone position therapy, encompassing the necessary hours and days in the prone position.

DETAILED DESCRIPTION:
The prone position leads to a more homogeneous distribution of ventilation by inflation of collapsed alveoli and reduction in alveolar hyperinflation. By employing EIT, the study can obtain a thorough comprehension of the ongoing alterations in regional ventilation before and after adopting the prone position. It is also anticipated that there is an impact on inflammation biomarkers before and after the prone position. This assessment aids in determining the ideal duration for prone position therapy, encompassing the necessary hours and days in the prone position.

Therefore, the investigators propose a project with the aim of collecting relevant clinical, laboratory, imaging, and respiratory physiology data from consenting patients with ARDS within the study period. The objective is to analyze changes in biomarkers following prone position.

ELIGIBILITY:
Inclusion Criteria:

1. Acute respiratory distress syndrome
2. Age > 18
3. Serial arterial blood gas data：PaO2/FiO2 <150. The mechanical ventilator setting：FiO2>0.6, PEEP>5 cmH2O

Exclusion Criteria:

1. Implantable electronic devices (e.g., pacemakers)
2. Body mass index > 30
3. Major thoracic and abdominal surgery
4. Patients with unstable spine and pelvis conditions
5. Pregnant women in the second and third trimesters
6. Patients with head trauma, elevated intracranial pressure, or elevated intraocular pressure
7. Hemodynamically unstable patients unsuitable for prone ventilation therapy
8. Patients with active seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focuses on patients with severe acute respiratory distress syndrome undergoing prone position therapy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prone response | During the prone position(5 days)
  Responder is defined as an increase in PaO2 by 20 mmHg or an increase in PaO2/FiO2 by 20% one hour after receiving prone position therapy

SECONDARY OUTCOMES:
28-day mortality | On the 28th day
  The mortality status on the 28th day

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yu Liao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No